CLINICAL TRIAL: NCT02810704
Title: Comparative Effectiveness of Pulmonary Embolism Prevention After Hip and Knee Replacement: Balancing Safety and Effectiveness
Brief Title: Comparative Effectiveness of Pulmonary Embolism Prevention After Hip and Knee Replacement
Acronym: PEPPER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Maryland, Baltimore (Other); Brigham and Women's Hospital (Other); Northwestern University (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Vincent D. Pellegrini, Professor of Orthopaedics, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FED19132
Record Dates: First submitted 2016-05-11; First posted 2016-06-23 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Embolism; Venous Thrombosis
Keywords: Anticoagulant; Venous Thromboembolism; Pulmonary Embolism; Total Knee Arthroplasty; Total Hip Arthroplasty
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Venous Thromboembolism | interventions — Aspirin; Warfarin; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Enteric Coated Aspirin (Experimental): Enteric coated aspirin (162 mg po) will be administered on the day of operation, prior to surgery, with a sip of water. Thereafter, starting on postoperative day #1, all patients in the aspirin group will receive 81 mg po bid to complete the treatment period of 30 days. Patients on preoperative cardiac dose aspirin may continue their usual dosing regimen prior to the morning of surgery, and then commence the PEPPER trial aspirin dose of 81 mg po bid on the day after operation.
  Interventions: Drug: Enteric Coated Aspirin
- Arm 2: Warfarin Other Names: Coumadin (Experimental): Warfarin will be administered starting on the day of operation, prior to surgery, with a sip of water. The initial dose will be empirically determined by body weight: less than 125 lbs (56.7 kg) - 2.5 mg; 125-250 lbs (56.7-113.4 kg) - 5 mg; greater than 250 lbs (113.4 kg) - 7.5mg. The initial dose will be repeated on the evening of surgery if the preoperative dose was administered prior to noon on the day of operation; no warfarin will be given on the evening of surgery if the preoperative dose was received after noon on the day of operation. Thereafter, starting on postoperative day #1, warfarin will be given each evening based on INR values to achieve a target of 2.0 (range 1.7-2.2).
  Interventions: Drug: Warfarin
- Arm 3: Rivaroxaban Other Names: Xarelto (Experimental): Rivaroxaban 10 mg will be first administered approximately 24 hours after completion of the index operation. Medication will then be administered in the evening on postoperative day #2 and thereafter each evening until completion.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Enteric Coated Aspirin
  Other Names: Aspirin
  Arms: Arm 1: Enteric Coated Aspirin
Drug: Warfarin
  Other Names: Coumadin
  Arms: Arm 2: Warfarin Other Names: Coumadin
Drug: Rivaroxaban
  Other Names: Xarelto
  Arms: Arm 3: Rivaroxaban Other Names: Xarelto

SUMMARY:
PEPPER is a randomized study comparing the three most commonly used anticoagulants in North America in patients who have elected to undergo primary or revision hip or knee joint replacement surgery. The anticoagulants being compared are enteric coated aspirin, low intensity warfarin, and rivaroxaban.

DETAILED DESCRIPTION:
PEPPER is a large pragmatic clinical trial to inform patient choice and balance risk tolerances of individuals who face decisions about different drugs and strategies for deep vein thrombosis (DVT) and pulmonary embolism (PE) prevention after total hip (THA) and knee (TKA) replacement. Indeed, clinical equipoise exists to ethically support such a randomized trial that has great potential to change current practice. We have selected the three prophylaxis methods that represent current orthopaedic practice in North America and collectively account for more than 80% of all hip and knee replacements; a) enteric coated aspirin (regimen with lowest bleeding risk; clinical PE and all-cause mortality rates comparable to more intensive anticoagulants), b) low intensity (INR Target 2.0) warfarin (time honored and one of the most common North American regimens; low bleeding risk [1-2%]), and c) rivaroxaban, a new oral direct Factor Xa inhibitor (regimen with lowest PE and DVT rate but higher bleeding risk [3-5%]). Prophylaxis will continue for 30 days, in accordance with clinical guidelines, and pneumatic compression will be utilized in hospital in conjunction with each treatment group. Each regimen is commonly used in contemporary practice, supported by observational and clinical trial data, and endorsed by the American College of Chest Physicians (ACCP) and American Academy of Orthopaedic Surgeons (AAOS) guidelines

ELIGIBILITY:
Inclusion Criteria:

1. 21 years of age or older;
2. Undergoing elective primary, revision or second stage re-implantation total hip/knee replacement or uni-compartmental knee replacement or hip resurfacing arthroplasty;
3. Has necessary mental capacity to participate and is able to comply with study protocol requirements;
4. Eligible for randomization to at least two of the three study regimens;
5. Is not pregnant on the day of surgery;
6. Has signed the consent form; and
7. Is willing to be randomized and participate in the study.

Exclusion Criteria:

1. Undergoing bilateral hip or knee replacement;
2. Has been previously enrolled;
3. Is pregnant or breastfeeding;
4. Is on chronic anticoagulation other than antiplatelet medications;
5. Concurrently enrolled in another active interventional clinical trial testing a drug or intervention known or believed to interact with aspirin, warfarin, or rivaroxaban;
6. Has documented gastrointestinal, cerebral, or other hemorrhage within 3 months;
7. Has a known diagnosis of defective hemostasis and past history of clinical bleeding requiring transfusion and treatment;
8. Has had an operative procedure involving the eye, ear, or central nervous system within one month;
9. Has uncontrolled hypertension with systolic BP > 220mmHg or diastolic BP > 120mmHg;
10. Body weight of less than 41 kilograms at baseline visit;
11. Member of a vulnerable patient population.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18883 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2025-09 (Actual); Study Completion 2025-09 (Actual)

PRIMARY OUTCOMES:
Aggregate primary clinical endpoints of all-cause mortality plus PE and DVT | Within 6 months of operation
  To compare the frequency of the aggregate primary clinical endpoints of important venous thromboembolism (clinical PE and DVT leading to hospital readmission) and all-cause mortality (aggregate indicator of fatal events, including both PE and major hemorrhage related to anticoagulant use) among three different venous thromboembolism (VTE) prophylaxis regimens. An audit of all hospital readmissions within 6 months of operation will be accomplished by routine postoperative follow-up through a mechanism of central telephone surveillance of patient-reported outcome events that is augmented by on-site research coordinator follow-up and validation of suspected endpoint events and adverse outcomes.
The frequency and nature of bleeding complications | Within 6 months of operation
  To compare the frequency and nature of bleeding complications (major, clinically important, and wound-related) leading to wound drainage, reoperation, or deep infection, or myocardial infarction among three different VTE prophylaxis regimens.
Specific Joint Function | Within 6 months of operation
  To compare the groups with respect to patient-reported outcomes in order to assess their impact on specific function of the replaced joint. Validated functional outcome tools will be compared among patients with and without primary endpoint events, as well as with historical baseline data warehoused in the FORCE registry, a national Agency for Healthcare Research and Quality (AHRQ) funded joint replacement outcomes database. Study site overlap with the FORCE registry is planned.
Patient Well- Being | Within 6 months of operation
  To compare the groups with respect to patient-reported outcomes in order to assess their impact on general patient well-being. Validated functional outcome tools will be compared among patients with and without primary endpoint events, as well as with historical baseline data warehoused in the FORCE registry, a national AHRQ funded joint replacement outcomes database. Study site overlap with the FORCE registry is planned.

SECONDARY OUTCOMES:
"Standard of care" methods of anesthesia on clinical effectiveness of three different prophylaxis regimens based on adverse events | Within 6 months of operation
  Analysis of the contribution of "standard of care" methods of anesthesia on clinical effectiveness of three different prophylaxis regimens. Stratification and subgroup analysis between patients with general compared with regional neuraxial (spinal/epidural) anesthesia will assess contribution of anesthesia to efficacy of VTE prophylaxis.
Comparative frequency of thromboembolic events and bleeding complications occurring after hip and knee replacement | Within 6 months of operation
  Analysis of the the relative frequency of thromboembolic events and bleeding complications in total hip compared with knee replacement patients. Evidence suggests etiology of venous thromboembolic disease (VTED) differs between THA and TKA and each may warrant a distinctive prophylaxis regimen based on likely outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent D Pellegrini, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Carol A Lambourne, PhD, Study Director — Dartmouth-Hitchcock Medical Center
Locations (32):
- United States (30):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA, Los Angeles, California
  - Stanford University Hospital, Stanford, California
  - Arthritis Surgery Research Foundation, South Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Sinai Hospital, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York University, New York, New York
  - Northwell Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Hershey Med Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Lifespan Health, East Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah
  - Anderson Orthopaedic Institute (VA), Alexandria, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The participating institutions will follow NIH guidelines concerning the sharing of research data. As outlined by the NIH and Patient-Centered Outcomes Research Institute (PCORI), the participating institutions will make available to the public the results of this collaboration and any accompanying data that were supported by PCORI. There are no specimens or biological resources for sharing as a result of this planned project.
  In the course of this research project, we anticipate generating ranges of estimated complications and adverse events as they relate to the use of VTE prophylaxis in the context of hip and knee replacement. Access to these data and associated recommendations generated under the project will be available for educational, research and non-profit purposes. Such access will be provided using web-based applications, as appropriate and consistent with the data distribution policies of the Medical University of South Carolina and the University of Maryland.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Spring 2024
Access Criteria: to be determined

REFERENCES:
- [Background] Pellegrini VD Jr, Eikelboom J, McCollister Evarts C, Franklin PD, Goldhaber SZ, Iorio R, Lambourne CA, Magaziner JS, Magder LS; Steering Committee of The PEPPER Trial. Selection Bias, Orthopaedic Style: Knowing What We Don't Know About Aspirin. J Bone Joint Surg Am. 2020 Apr 1;102(7):631-633. doi: 10.2106/JBJS.19.01135. No abstract available. PMID 31895235
- [Background] Pellegrini VD Jr, Eikelboom JW, Evarts CM, Franklin PD, Garvin KL, Goldhaber SZ, Iorio R, Lambourne CA, Magaziner J, Magder L; Steering Committee of the PEPPER Trial and the PEPPER Trial Investigators, funded by PCORI. Randomised comparative effectiveness trial of Pulmonary Embolism Prevention after hiP and kneE Replacement (PEPPER): the PEPPER trial protocol. BMJ Open. 2022 Mar 8;12(3):e060000. doi: 10.1136/bmjopen-2021-060000. PMID 35260464
- [Derived] Hanson TM, Magder LS, Pellegrini VD Jr; PEPPER Trial Investigators. Substantial Improvement in Self-Reported Mental Health Following Total Hip Arthroplasty Occurs Independent of Anesthetic Technique. J Arthroplasty. 2024 May;39(5):1220-1225.e1. doi: 10.1016/j.arth.2023.11.011. Epub 2023 Nov 17. PMID 37977307
- [Derived] Ko H, Pelt CE, Martin BI; PEPPER Investigators; Pellegrini VD Jr. Patient-reported outcomes following cemented versus cementless primary total knee arthroplasty: a comparative analysis based on propensity score matching. BMC Musculoskelet Disord. 2022 Oct 27;23(1):934. doi: 10.1186/s12891-022-05899-1. PMID 36303136
- [Derived] Finch DJ, Martin BI, Franklin PD, Magder LS, Pellegrini VD Jr; PEPPER Investigators. Patient-Reported Outcomes Following Total Hip Arthroplasty: A Multicenter Comparison Based on Surgical Approaches. J Arthroplasty. 2020 Apr;35(4):1029-1035.e3. doi: 10.1016/j.arth.2019.10.017. Epub 2019 Oct 17. PMID 31926776